CLINICAL TRIAL: NCT03192098
Title: Progressive Versus Conservative Dilation Strategy for Benign Esophageal Strictures: a Randomized Controlled Trial
Brief Title: Progressive Esophageal Dilation for Benign Strictures: a Randomized Controlled Trial
Acronym: DILATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL.60222.901.16
Record Dates: First submitted 2017-05-29; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Benign Esophageal Stricture

STUDY DESIGN:
Intervention Model Description: randomized controlled patient groups
Who Masked: Participant
Masking Description: Participant will be blinded for dilation strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive (Experimental): Patients will be dilated > 3mm and can be dilated up to 6mm in diameter
  Interventions: Device: Savary bougie dilation
- Conservative (rule-of-3) (Active Comparator): Patients will be dilated according to the rule-of-3 (i.e. dilation of no more than 3mm in diameter)
  Interventions: Device: Savary bougie dilation

INTERVENTIONS:
Device: Savary bougie dilation — Patients will be dilated with the use of the Savary bougienage device

SUMMARY:
A randomized controlled prospective clinical trial assessing the efficacy and safety of progressive esophageal dilation compared to conservative esophageal dilation in patients with severe benign esophageal strictures.

DETAILED DESCRIPTION:
A randomized controlled prospective clinical trial assessing the efficacy and safety of progressive esophageal dilation (up to 6mm) compared to esophageal dilation according to the rule-of-3 in patients with severe benign esophageal strictures. Patients will be followed up for 6 months. When recurrent dysphagia occurs within 6 months the patients will be dilated according to the previously allocated strategy.

ELIGIBILITY:
Inclusion Criteria:

* Dysphagia due to benign esophageal stricture (e.g. surgery, radiation therapy, caustic ingestion, peptic injury, photodynamic therapy) requiring esophageal dilation
* Requiring first esophageal dilation for dysphagia due to a severe benign esophageal stricture with no patency for standard upper endoscope (9-10mm diameter)
* No history of esophageal endoscopic dilations for benign strictures the past 6 months
* Dysphagia for solid, semisolid or liquid food (dysphagia score ≥ 2 [Ogilvie]16, and dysphagia score ≤ 21 [Dakkak and Bennett]19, see appendix)
* Written informed consent

Exclusion Criteria:

* Patient < 18 years old
* Patient is unwilling or unable to sign and date the informed consent
* Patient is unwilling or unable to comply with the follow-up schedule
* Patient is unable to understand informed consent and fill in the questionnaires due to a language barrier
* Patient is pregnant, breast-feeding, or planning to become pregnant in the next 12 month
* Patient is simultaneously participating in another drug or device study or the patient has completed the follow-up phase for the primary objective of any previous study less than 30 days prior to enrollment in this study
* Previous esophageal dilation for benign stricture within the past 6 months
* Patient with a life expectancy < 12 months
* Patient with a known eosinophilic esophagitis or motility disorder (such as achalasia)
* Patients with a known malignant esophageal stricture
* Patients with a benign stricture due to a previous performed laryngectomy

Endoscopic exclusion criteria:

* Benign strictures in the upper part of the esophagus too close to the cricopharyngeal muscle (for the purpose of this protocol, within 1½ cm of the upper esophageal sphincter)
* Patients with stricture ≥ 10 cm in length
* Patients with an active esophageal perforation, leak, fistula, or varices
* Stricture within necrotic chronically bleeding tumors
* Highly suspected esophageal malignancy
* Stricture within polypoid lesions
* Known or strongly suspected dysmotility esophageal disorder
* Patient with high suspicion for an esophageal web, Schatzki ring, eosinophilic esophagitis, or motility disorder (such as achalasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Total number of dilation procedures within 6 months of follow-up | 6 months
  Total number of dilation procedures within 6 months of follow-up
Total number of dilation procedures during first dilation session to 16-18mm | 1 month
  Total number of dilation procedures during first dilation session to 16-18mm

SECONDARY OUTCOMES:
Dysphagia free patients | 6 months
  Number of patients remaining dysphagia free within 6 months after dilation to 16-18mm
Timeframe first dilation session | 1 month
  Time from first dilation session to dilation of 16-18mm
Dysphagia free time period | 6 months
  Time to dilation of recurrent stricture after initial dilation to 16-18mm
Incidence of treatment-related mortality (serious) adverse events (safety) | 7 months
  Incidence of treatment-related mortality (serious) adverse events (safety)
Quality of Life | 6 months
  SF-36, disease specific questionnaire
Medical costs | 7 months
  Direct medicals costs: procedures, secondary interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No